CLINICAL TRIAL: NCT00117390
Title: Evaluation of the Optimal Technique for Determination of the Renal Function of Critically Ill Patients
Brief Title: Evaluation of the Optimal Technique for Determination of Renal Function of Critically Ill Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Ghent (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2004/101
Record Dates: First submitted 2005-06-30; First posted 2005-07-06 (Estimated); Last update posted 2007-12-28 (Estimated); Status verified 2007-12

CONDITIONS: Renal Function; Critical Illness
MeSH Terms: conditions — Critical Illness

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Measurement of inulin clearance

SUMMARY:
The purpose of this study is to evaluate the optimal technique for determination of the renal function of critically ill patients.

ELIGIBILITY:
Inclusion Criteria:

* Over 18 years old
* Intensive care patient
* Given informed consent
* Arterial infusion
* A bladder catheter

Exclusion Criteria:

* Diurese < 400 mL/d

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50
Dates: Start 2004-06; Study Completion 2006-10 (Actual)

PRIMARY OUTCOMES:
Comparison of the determination of the renal function by other means than the golden standard, inulin clearance

CONTACTS AND LOCATIONS:
Overall Officials: Eric Hoste, MD, PhD, Principal Investigator — University Hospital, Ghent
Locations (1):
- University Hospital Ghent, Ghent, Belgium

REFERENCES:
- See also: Website of the University Hospital Ghent — http://www.uzgent.be